CLINICAL TRIAL: NCT00120510
Title: A Randomized Clinical Trial to Determine the Efficacy of Early Versus Standard Antiretroviral Therapy in HIV Infected Adults With CD4+ T Cell Counts Between 200 and 350 Cells/mm3
Brief Title: Early Versus Standard Start of Anti-HIV Therapy for Treatment-Naive Adults in Haiti
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIPRA HT 001; 5K24AI051966-03 (NIH); 10403 (Registry Identifier: DAIDS ES number)
Record Dates: First submitted 2005-07-14; First posted 2005-07-18 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: HIV Infections; Tuberculosis
Keywords: Treatment Naive; TB
MeSH Terms: conditions — HIV Infections; Tuberculosis | interventions — efavirenz; lamivudine, zidovudine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Randomly assigned group who will start an ART regimen of 3TC/ZDV and EFV twice daily at study entry
  Interventions: Drug: Efavirenz; Drug: Lamivudine/Zidovudine
- B (Active Comparator): Randomly assigned group who will delay beginning ART regimen of 3TC/ZDV and EFC twice daily until they develop clinical AIDS or their CD4 count drops below 200 cells/mm3
  Interventions: Drug: Efavirenz; Drug: Lamivudine/Zidovudine

INTERVENTIONS:
Drug: Efavirenz — Non-nucleoside reverse transcriptase inhibitor dosed at 600mg taken by mouth every 24 hours at bedtime
  Other Names: EFV
Drug: Lamivudine/Zidovudine — Nucleoside reverse transcriptase inhibitor dosed at 150mg/300mg fixed dose combination taken by mouth every 12 hours
  Other Names: 3TC/ZDV; 3TC/AZT

SUMMARY:
Anti-HIV treatment consisting of lamivudine/zidovudine (3TC/ZDV) and efavirenz (EFV) is the current standard of care for initial treatment of HIV in most areas of the world. The purpose of this study is to determine the best time to start this anti-HIV treatment in treatment-naive adults in Haiti.

DETAILED DESCRIPTION:
In many parts of the world, initial standard of care for HIV includes 3TC/ZDV and the non-nucleoside reverse transcriptase inhibitor EFV. However, it is unclear if early (CD4 count less than 350 cells/mm3) or delayed (CD4 count less than 200 cells/mm3) therapy initiation leads to improved survival. This study will determine the most appropriate time to initiate ART in HIV infected individuals in Haiti. The study will enroll patients from the Haitian Study Group on Kaposi's Sarcoma and Opportunistic Infections (GHESKIO) Centers. Some participants in this study will have active pulmonary tuberculosis (TB).

This study will last at least 3 years. Participants will be randomly assigned to one of two groups at study entry. Group A participants will receive 3TC/ZDV twice daily and EFV once daily at study enrollment. Participants receiving TB therapy at the time of enrollment may be observed for 2 weeks prior to beginning early therapy. Dosage adjustment of EFV may be necessary for participants receiving rifampin as part of their TB therapy. Group B participants will receive 3TC/ZDV twice daily and EFV once daily when they develop clinical AIDS or their CD4 count drops below 200 cells/mm3 (WHO Stage IV). Directly observed therapy will be used for the first two months of treatment for every participant.

Group A participants will have 14 study visits after beginning treatment; the visits will occur at Months 1, 2, 3, and every 3 months thereafter. Medical and medication history, physical exams, and contraceptive counseling for women will occur at all visits. HIV counseling, blood collection, and HIV staging will occur at most visits. At some study visits, Group A participants will be asked to complete quality of life and adherence questionnaires. Group B participants will have 14 study visits after study entry and will begin treatment when they meet WHO criteria. Assessments will be the same as for Group A. Any participant who fails the first-line regimen during the study will switch to a second-line ART regimen.

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected
* Received pre- and post-test counseling at the GHESKIO Centers
* CD4 count between 200 and 350 cells/mm3
* World Health Organization (WHO) Stage I, II, or III HIV disease
* Willing to use acceptable forms of contraception

Exclusion Criteria:

* WHO Stage IV HIV disease (AIDS)
* 7 or more days of cumulative ART prior to study entry OR on ART at time of study entry
* Active TB, if diagnostic work-up for TB is incomplete OR if decision to treat TB has not been made. More information on this criterion can be found in the protocol.
* Recurrent active TB OR history of interrupted or incomplete TB therapy. More information on this criterion can be found in the protocol.
* Has not been evaluated for latent TB and decision to treat latent TB with isoniazid has not been made. More information on this criterion can be found in the protocol.
* Requires ART in the next 3 months, in the opinion of the investigator
* Other serious medical illness requiring chronic maintenance therapy (e.g., hypertension, diabetes) UNLESS the individual has completed at least 14 days of therapy prior to study enrollment AND is clinically stable
* Any psychological condition (e.g., severe depression, schizophrenia) that, in the opinion of the investigator, may interfere with the study
* Any social condition (e.g., pending emigration, pending incarceration) that, in the opinion of the investigator, may interfere with the study
* Active drug or alcohol use that, in the opinion of the investigator, may interfere with the study
* Current inflammation of the pancreas
* Allergy/sensitivity to any of study drugs or their formulations
* Requires certain medications
* Enrolled in another therapeutic or interventional clinical trial
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 816 (Actual)
Dates: Start 2007-07; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Survival | At 36 months

SECONDARY OUTCOMES:
Safety and drug-associated side effects and toxicities of the study drugs | Throughout study
Pattern and frequency of antiretroviral drug resistance during ART | Throughout study
Occurrence and clinical outcome of opportunistic infections, viral coinfections, and immune reconstitution syndromes observed during ART | Throughout study
TB treatment outcomes in patients with active pulmonary TB at enrollment | Throughout study
Quality of life scores based on self-report questionnaires | Throughout study
Adherence based on self-report questionnaires and dosage count | Throughout study
Cost of therapy | Throughout study
Plasma HIV-1 RNA below limits of quantitation after initiating ART | Every 6 months throughout study
Absolute CD4 cell count change from baseline in subjects who initiate ART | Every 6 months throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Jean William Pape, MD, Principal Investigator — Cornell - GHESKIO, Institut de Laboratoire et de Recherches and Division of International Medicine and Infectious Diseases, Cornell University; Patrice Severe, MD, Study Director — Cornell - GHESKIO, Institut de Laboratoire et de Recherches; Daniel W. Fitzgerald, MD, Study Director — Division of International Medicine and Infectious Diseases, Cornell University
Locations (1):
- Les Centres GHESKIO CIPRA CRS, Port-au-Prince, Haiti

REFERENCES:
- [Background] Blankson JN. Primary HIV-1 infection: to treat or not to treat? AIDS Read. 2005 May;15(5):245-6, 249-51. PMID 15900634
- [Background] Duncombe C, Kerr SJ, Ruxrungtham K, Dore GJ, Law MG, Emery S, Lange JM, Phanuphak P, Cooper DA. HIV disease progression in a patient cohort treated via a clinical research network in a resource limited setting. AIDS. 2005 Jan 28;19(2):169-78. doi: 10.1097/00002030-200501280-00009. PMID 15668542
- [Background] Pape JW. Tuberculosis and HIV in the Caribbean: approaches to diagnosis, treatment, and prophylaxis. Top HIV Med. 2004 Dec-2005 Jan;12(5):144-9. PMID 15647610
- [Background] Teck R, Ascurra O, Gomani P, Manzi M, Pasulani O, Kusamale J, Salaniponi FM, Humblet P, Nunn P, Scano F, Harries AD, Zachariah R. WHO clinical staging of HIV infection and disease, tuberculosis and eligibility for antiretroviral treatment: relationship to CD4 lymphocyte counts. Int J Tuberc Lung Dis. 2005 Mar;9(3):258-62. PMID 15786887
- [Background] Thorner A, Rosenberg E. Early versus delayed antiretroviral therapy in patients with HIV infection : a review of the current guidelines from an immunological perspective. Drugs. 2003;63(13):1325-37. doi: 10.2165/00003495-200363130-00001. PMID 12825959
- [Derived] Joseph Y, Yao Z, Dua A, Severe P, Collins SE, Bang H, Antoine Jean-Juste M, Ocheretina O, Apollon A, McNairy ML, Dupnik K, Cremieux E, Byrne A, Pape JW, Koenig SP. Long-term mortality after tuberculosis treatment among persons living with HIV in Haiti. J Int AIDS Soc. 2021 Jul;24(7):e25721. doi: 10.1002/jia2.25721. PMID 34235862
- [Derived] Collins SE, Jean Juste MA, Koenig SP, Secours R, Ocheretina O, Bernard D, Riviere C, Calnan M, Dunning A, Hurtado Rua SM, Johnson WD Jr, Pape JW, Fitzgerald DW, Severe P. CD4 deficit and tuberculosis risk persist with delayed antiretroviral therapy: 5-year data from CIPRA HT-001. Int J Tuberc Lung Dis. 2015 Jan;19(1):50-7. doi: 10.5588/ijtld.14.0217. PMID 25519790
- [Derived] Haas DW, Severe P, Jean Juste MA, Pape JW, Fitzgerald DW. Functional CYP2B6 variants and virologic response to an efavirenz-containing regimen in Port-au-Prince, Haiti. J Antimicrob Chemother. 2014 Aug;69(8):2187-90. doi: 10.1093/jac/dku088. Epub 2014 Apr 2. PMID 24695352
- [Derived] Koenig SP, Bang H, Severe P, Jean Juste MA, Ambroise A, Edwards A, Hippolyte J, Fitzgerald DW, McGreevy J, Riviere C, Marcelin S, Secours R, Johnson WD, Pape JW, Schackman BR. Cost-effectiveness of early versus standard antiretroviral therapy in HIV-infected adults in Haiti. PLoS Med. 2011 Sep;8(9):e1001095. doi: 10.1371/journal.pmed.1001095. Epub 2011 Sep 20. PMID 21949643
- [Derived] Severe P, Juste MA, Ambroise A, Eliacin L, Marchand C, Apollon S, Edwards A, Bang H, Nicotera J, Godfrey C, Gulick RM, Johnson WD Jr, Pape JW, Fitzgerald DW. Early versus standard antiretroviral therapy for HIV-infected adults in Haiti. N Engl J Med. 2010 Jul 15;363(3):257-65. doi: 10.1056/NEJMoa0910370. PMID 20647201